CLINICAL TRIAL: NCT03598439
Title: Randomized Open-Label Trial to Compare Immunogenicity of Egg-Based and Non-Egg Based Quadrivalent Influenza Vaccines Among Adults 18-64 Years of Age (US Flu Vaccine Effectiveness Serologic Study, 2018-19 and 2019-20)
Brief Title: Randomized Influenza Vaccine Evaluation of Immune Response
Acronym: RIVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marshfield Clinic Research Foundation (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Huong Nguyen, PhD, Senior Research Scientist, Marshfield Clinic Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MCL10218
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Influenza
Keywords: influenza vaccine; adults; Immune response
MeSH Terms: conditions — Influenza, Human | interventions — Cell Culture Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Recombinant (RIV4) Influenza Vaccine (Experimental): A single dose of licensed recombinant influenza vaccine will be given in each of two influenza seasons - one in 2018-19 and a second in 2019-20.
  Interventions: Biological: Recombinant
- Cell-culture (ccIIV4) Influenza Vaccine (Experimental): A single dose of licensed cell-culture influenza vaccine will be given in each of two influenza seasons - one in 2018-19 and a second in 2019-20
  Interventions: Biological: Cell-culture
- Standard (IIV4) Influenza Vaccine (Active Comparator): A single dose of licensed standard influenza vaccine will be given in each of two influenza seasons - one in 2018-19 and a second in 2019-20.
  Interventions: Biological: Standard IIV4

INTERVENTIONS:
Biological: Standard IIV4 — Standard inactivated influenza vaccine
  Other Names: Flulaval Quadrivalent
  Arms: Standard (IIV4) Influenza Vaccine
Biological: Recombinant — Influenza vaccine that uses a hemagglutinin protein manufactured in insect cells with a baculovirus vector
  Other Names: FluBlok Quadrivalent
  Arms: Recombinant (RIV4) Influenza Vaccine
Biological: Cell-culture — inactivated influenza vaccine manufactured using mammalian cell lines; current vaccine uses a cell-propagated H3N2 strain.
  Other Names: Flucelvax Quadrivalent
  Arms: Cell-culture (ccIIV4) Influenza Vaccine

SUMMARY:
Licensed influenza vaccines are manufactured with a variety of technologies. The majority are split, inactivated vaccines derived from egg-adapted, high growth reassortant viruses. Two US licensed products do not use egg-adapted viruses: Flucelvax (mammalian cell culture) and FluBlok (recombinant). There is increasing evidence that egg propagation induces virus mutations that impair the immune responses to circulating viruses. However, the impact of egg-propagation on clinical vaccine effectiveness is uncertain, and there is no preferential recommendation for any specific influenza vaccine product or technology. A direct comparison of serologic response to egg based and non-egg based vaccines in adults has not been performed. This randomized trial will compare serologic responses to the egg- and non-egg A(H3N2) vaccine component. The study cohort will be followed for two influenza seasons to evaluate sequential vaccination effects on immune response.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-64 years
* Marshfield Clinic patients living in or around Marshfield, Wisconsin since July 2015
* Willing and able to give informed consent and comply with study requirements

Exclusion Criteria:

* Receipt of 2018-19 influenza vaccine prior to study enrollment
* Known to be pregnant at the time of enrollment
* Current participation or plans to participate in another clinical trial involving an experimental agent
* Presence of a contraindication to influenza vaccination
* Plans to relocate outside the geographic location in the next two years

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 366 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Post-vaccination titer | 28 days
  geometric mean titers (as measured by microneutralization) to cell-grown A(H3N2) vaccine reference virus

CONTACTS AND LOCATIONS:
Locations (1):
- Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No